CLINICAL TRIAL: NCT01299246
Title: The Effectiveness of Improving Self-care and Health Status After Promoting Counseling for the Diabetics Mellitus Patients With DM Foots Around Yunlin and Chiayi Region
Brief Title: The Effectiveness of Improving Self-care After Counseling for the Diabetics Mellitus Foots Around Chiayi Region
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Chang Gung Memorial Hospital, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Screening
Other Study IDs: 98-2224-B
Record Dates: First submitted 2011-01-30; First posted 2011-02-18 (Estimated); Last update posted 2011-02-18 (Estimated); Status verified 2009-10

CONDITIONS: Diabetic Foot; Type 2 Diabetes Mellitus With Established Diabetic Nephropathy
Keywords: Diabetic Foot; non-invasive DFP assessment tools; early detection of DFP
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- improving self-care (Experimental)
  Interventions: Procedure: Michigan Neuropathy Screening Instrument

INTERVENTIONS:
Procedure: Michigan Neuropathy Screening Instrument — Peripheral neurological assessment was carried out using MNSI. The diabetes nurse educators assessed five parameters on both feet and counted the total points, ranging from 0 to10: (1) Appearance of feet; if abnormal, then inspection of lower limbs for deformities was carried out; (2) Identification of foot ulceration; (3) Vibration perception of the big toe; (4) Ankle reflexes; (5) touch-pressure sensation test with a 10 g Semmes-Weinstein monofilament.
  Other Names: Cardio-Vision Model MS-2000 for ABI measurement.

SUMMARY:
Objectives:

Preventing diabetic foot problems (DFP) and associated consequences, such as amputation, is a critical in rural regions. The objective is to present on the association of non-invasive DFP assessment tools and physiological indicators for the early detection of DFP among rural cases of diabetes in Taiwan.

DETAILED DESCRIPTION:
1. Peripheral neurological assessment was carried out using Michigan Neuropathy Screening Instrument (MNSI). The diabetes nurse educators assessed five parameters on both feet and counted the total points, ranging from 0 to10: (1) Appearance of feet (normal/abnormal with 0 and 1 point); if abnormal, then inspection of lower limbs for deformities, dry skin, fissure, calluses or infection was carried out; (2) Identification of foot ulceration (yes/no with 0 and 1 point); (3) Vibration perception of the big toe (present/decreased/absent, with 0, 0,5 and 1 points); (4) Ankle reflexes (present/reinforcement/absent, with 0, 0,5 and 1 points); (5) touch-pressure sensation test with a 10 g Semmes-Weinstein monofilament (normal/reduced/absent, with 0, 0,5 and 1 points). When an MNSI summative score was ≥2 points with neuropathy, patients were referred to the teaching hospitals for further evaluation. The MNSI procedures took 6-8 minutes for each participant.
2. Peripheral vascular assessment: three parameters were used to assess peripheral vascular function by trained nurses. (a) The Cardio-Vision Model MS-2000 was used to detect Ankle Brachial Index (ABI), assessed by research nurses. Values of ABI were classified as ≥0.9 normal and <0.9 abnormal. (b) Palpable pedal, posterior tibias and popliteal pulses were recorded as absent, weak or present. (c) Capillary refill time was done by pressing the tip of the toenail for two seconds, and taking the time for the blanched area to turn pink again. If the return time took >2 seconds, this was taken as ischemia. Assessing of all 3 parameters of peripheral vascular assessment took 10-15 minutes for each participant.
3. Diabetic foot risk assessment was assessed by plastic surgeons: (a) King's College classification (KC) contained six stages of condition: not at risk, at risk, ulcer, cellulites, necrosis and amputation. (b) the Texas risk classification (TRC) system was divided into six categories in origin. We re-categorized three levels: low risk, at risk, and high risk.
4. The blood glucose, total cholesterol, and low density of lipoprotein cholesterol were drawn from the last 1-2 month diabetes passport record for each subject. Blood pressure was measured according to standard procedures by the nurses during the study. Body mass index was calculated for each participant using the standard formula (weight in kilograms divided by square of the height in meters). Waist circumference in centimeter was used to measure central obesity, measuring the mid-abdominal distance between the last rib margin and the iliac crest.

ELIGIBILITY:
Inclusion Criteria:

* diabetics mellitus patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 386 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Number of the residents in detecting the early neurovasculopathy | 1 year
  It is shown that using the MNSI and ABI as community screening tools can be useful in detecting the early neurovasculopathy for diabetic rural residents. In addition, where an ABI machine is unavailable, performing MNSI using primary healthcare providers might be cost-effective.

CONTACTS AND LOCATIONS:
Overall Officials: Mei-Yen Chen, Ph.D., Study Chair — Graduate Institute of Nursing, Chang Gung Institute of Technology, Chiayi Campus, Taiwan. Tel: 886 (5) 3628800 ext. 2201, Fax: 886-5-3628866, Email: meiyen@gw.cgit.edu.tw
Locations (1):
- Graduate Institute of Nursing, Chang Gung Institute of Technology, Chiayi Campus, Chiayi City, Taiwan